CLINICAL TRIAL: NCT03331146
Title: Randomized, Controlled, Double-blinded Pilot Study: Nitrite Infusion in High Risk Patients Undergoing Cardiopulmonary Bypass
Brief Title: Nitrite Infusion in High Risk Patients Undergoing Cardiopulmonary Bypass
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Principal Investigator made aware of similar studies that have already been published.
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Ahmed Zaky, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 1709284471
Record Dates: First submitted 2017-10-20; First posted 2017-11-06 (Actual); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Acute Kidney Injury
Keywords: Nitric Oxide; Sodium Nitrite; Cardiopulmonary bypass; cardioplegic cardiac arrest; coronary revacularization
MeSH Terms: conditions — Acute Kidney Injury | interventions — Sodium Chloride; Sodium Nitrite

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control group (Placebo Comparator): saline infusion will be administered after induction of general anesthesia
  Interventions: Drug: Saline; Drug: Sodium Nitrite
- Sodium Nitrite (Active Comparator): sodium nitrite will start after induction of general anesthesia via a dedicated IV line for 6 hrs.
  Interventions: Drug: Saline; Drug: Sodium Nitrite

INTERVENTIONS:
Drug: Saline — A placebo (saline infusion) will be administered after induction of general anesthesia.
Drug: Sodium Nitrite — Sodium nitrite infusion at a 267 mcg/kg/hr. will start after induction of general anesthesia via a dedicated IV line for 6 hrs.
  Other Names: NaNO2

SUMMARY:
The main objective of this study is to evaluate the efficacy of intravenous sodium nitrite compared with placebo in reducing the occurrence of CSA-AK as diagnosed by KDIGO criteria during the first 72 hrs after cardiac surgery in high-risk patients undergoing cardiac surgery. Secondary objectives are to determine whether IV sodium nitrite achieves adequate pharmacokinetics (PK) in patients undergoing cardiac surgery with the use of CPB.

DETAILED DESCRIPTION:
Acute kidney injury is one of the most untoward consequences of cardiac-surgery with the use of CPB. As such it is associated with a high mortality and morbidity and health care expense. Unfortunately, currently, there is no effective preventive or treatment strategy for cardiac surgery-associated (CSA) AKI other than renal replacement therapy.

It is postulated that a major mechanism of CSA-AKI is created by the ischemia reperfusion injury (IRI) resulting from aortic cross clamping and unclamping. This creates a cascade of events culminating in inflammation, microvascular dysfunction and tubular cell maladaptation and eventually renal tissue damage. Current treatment modalities that target the microcirculation such as blood pressure and cardiac output fails to prevent renal abnormalities and as such may be deleterious to the renal tissue microcirculation. The PI hypothesizes that a therapeutic strategy that limits IRI such as the administration of inhaled nitric oxide (NO) or sodium nitrite (NaNO2) would ameliorate CSA-AKI by limiting inflammatory injury to the kidney.

The anion nitrite (NO2-) releases NO in biological systems and has been demonstrated to inhibit IR injury in the heart, liver and kidneys created by various pathologic states1-3 and improve outcomes in patients with acute myocardial infarction, in patients with pulmonary hypertension and is the putative active mediator of protection in liver-transplantation patients receiving inhaled nitric oxide4.

The objective of this study is to determine whether the NO donor, nitrite will prevent I/R injury in patients at high risk of development of CSA-AKI undergoing open-heart surgery with cardiopulmonary bypass.

ELIGIBILITY:
Inclusion Criteria:

* Patients CCFS score ≥ 6 (Table 1)
* Patients admitted to UAB cardiac intensive care unit (CICU) following elective cardiac surgery with cardiopulmonary bypass under general endotracheal anesthesia
* 19 years old
* Estimated glomerular filtration rate (eGFR) ≥ 30 ml/min/1.73 m2

Exclusion Criteria:

* Prisoners directly admitted from a correctional facility.
* Children < 19 years or under 50 kg body weight if age is unknown.
* Patients enrolled in a concurrent ongoing interventional, randomized clinical trial.
* Patients with end stage renal disease or preexisting GFR <30 mL/min/1.73 m2 or need for dialysis. 34
* Patients with end stage heart disease on the cardiac transplant list.
* Patients undergoing procedures without the use of CPB
* All transplant patients.
* Patients on ventricular assist devices.
* Patients undergoing emergency procedures.
* Patients with glucose 6-dehydrogenase deficiency
* Pregnancy

Ages: 19 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2019-06-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Nitrite Metabolome Levels | baseline to 73 hrs post-operatively
  Measuring nitrite, nitrate, and nitrosothiols levels
Biomarkers of Hemolysis | baseline to 73 hrs post-operatively
  Measuring hemolysis indicators heme, Hb, hemopexin, and hemopectin
Biomarkers of Kidney Injury | baseline to 73 hrs post-operatively
  Measuring kidney injury indicators creatine, neutrophil-associated gelatinase, lipocalin (NGAL)
Cell Cycle Stress | baseline to 73 hrs post-operatively
  Measuring cell cycle arrest biomarkers TIMP-2, IGFBP-7

SECONDARY OUTCOMES:
Biomarkers of Hepatic injury | baseline to 24 hours post-operatively
  Measuring serum AST and ALT
Biomarkers of Kidney Injury | baseline to 24 hours post-operatively
  Measuring kidney injury indicators creatine, neutrophil, lipocalin (NGAL)
Cell Cycle Stress | baseline to 24 hours post-operatively
  Measuring cell cycle arrest biomarkers TIMP-2, IGFBP-7
Biomarkers of Myocardial Injury | baseline to 24 hours post-operatively
  Measuring myocardial injury indicators troponin and CKMB
Urine Output | baseline to 73 hrs post-operatively
  Measuring total urine output
Vasopressors Usage | baseline to 73 hrs post-operatively
  Percentage of vasopressor usage between the control and intervention

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed F Zaky, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB Department of Anesthesiology and Perioperative Medicine, Birmingham, Alabama, United States